CLINICAL TRIAL: NCT05817578
Title: Profiling the Rotator Cuff - Related Shoulder Pain (RCRSP) Patient: a Pain Phenotype Classification Algorithm
Brief Title: Profiling the RCRSP Patient: a Pain Phenotype Classification Algorithm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Achilleas Paliouras, Principal Investigator, Physiotherapist, MSc, PhD candidate, University of Thessaly
Other Study IDs: 9
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Rotator Cuff Syndrome; Rotator Cuff Tears; Rotator Cuff Tendinosis; Rotator Cuff Impingement; Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: Rotator Cuff Related Shoulder Pain; Chronic Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome; Rupture; Chronic Pain | interventions — Arthrometry, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Quantitative Sensory Testing / Dynamometry / Goniometry — Testing procedures that follow previously used protocols of the literature for all the Quantitative Sensory Testing, Dynamometry & Goniometry
  Other Names: Dynamometry; Goniometry

SUMMARY:
The aim of this study is to collect a sum of different characteristics that have been mentioned previously in people presenting with RCRSP and by clustering them to create a phenotype system which may assist the individualisation of their management

DETAILED DESCRIPTION:
This study will be conducted at a hospital environment by recruiting people that will seek help for their shoulder pain by a specialist upper- limb Orthopaedic Surgeon at the Department of Hand & Upper Limb Microsurgery of the 'KAT General Hospital' in Athens, Greece. Participants that will be diagnosed with RCRSP by the orthopaedic surgeon and fulfil the eligibility criteria will undergo a series of one-off measurements. Written consent will have to be obtained before a sum of self-reported outcome measures and objective testing will take place. The main categories for which outcome measures will be used are: pain, function, psychosocial and lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* Pain: >3 months, non-traumatic, unilateral or bilateral of anterolateral location
* ROM: >50% all planes, AROM painful in forward flexion and/or abduction
* Provocation testing: Hawkins-Kennedy, Neer, Painful Arc, Resisted ER, Empty Can (3 or more out of the 5 +ve)

Exclusion Criteria:

* Pain < 3months
* History of neck or shoulder trauma
* Radicular signs, shoulder pain reproduced with neck movements
* GH OA
* Frozen Shoulder
* Tears >C3 according to Snyder Classification
* Fibromyalgia
* Neurological, systemic local or autoimmune inflammatory conditions
* Clinical depression
* No injected corticosteroids or physiotherapy the last 3/12

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People in the 18-65 spectrum that have a gradual onset of shoulder pain without being able to recall any injuries to the area and pain to be present for at least three months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-02 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Once - Baseline
  Obtain a measurement of pain
  Score: 0-10
  Higher scores indicate more pain
Western Ontario Rotator Cuff Index (WORC) | Once - Baseline
  Assess the self-reported functional ability of participants
  Score: 0-100 %
  Higher scores indicate higher functional status
The Self-Report Leeds Assessment of Neuropathic Symptoms & Signs (SLANSS) | Once - Baseline
  Identify possible participants with neuropathic type of pain
  Score: 0-24
  Score >12 indicates neuropathic pain
Central Sensitisation Inventory (CSI) | Once - Baseline
  Identify participants suspicious of central sensitisation symptoms
  Score: 0-100
  Score>40 indicates central sensitisation
Pain Drawings (PD) | Once - Baseline
  Capture painful body locations for participants with the spectrum of pathologies
Nociplastic Pain Flow Chart by IASP | Once - Baseline
  Identification of Predominant Pain Mechanism, especially participants with possible nociplastic pain
Quantitative Sensory Testing (QST) | Once - Baseline
  Assessment of Pressure Pain Threshold, Conditioned Pain Modulation & Temporal Summation
Range of Motion (ROM) | Once - Baseline
  Assess Range of motion of the movements of interest
Dynamometry | Once - Baseline
  Assess strength and explore pain provocation in participants
Posterior Shoulder Endurance Test (PSET) | Once - Baseline
  Assess the endurance of the Rotator Cuff myotendinous unit
Hospital Anxiety & Depression Scale (HADS) | Once - Baseline
  Obtain a score of Anxiety & Depression among participants
  Score: 0-42 (Two scales between 0 & 21 each - one for anxiety and 1 for depression)
  Higher Scores indicate higher anxiety & depression
Pain Catastrophising Scale (PCS) | Once - Baseline
  Explore how the pain experience is perceived by the individual
  Scale: 0-52
  Higher scores indicate higher levels of catastrophising
Tampa Scale of Kinesiophobia (TSK) | Once - Baseline
  Explore fear of movement and avoidance of participants
  Score: 17-68
  Higher scores indicate higher levels of Kinesiophobia, cut-off point: scores >37 are indicative of kinesiophobia
Pain Self-Efficacy Questionnaire (PSEQ) | Once - Baseline
  Assess the ability of the participant to cope with a spectrum of activities
  Score: 0-60
  Lower scores indicate less self-efficacy
Allostatic Index-5 (ALI-5) | Once - Baseline
  Investigate psychosocial stressors reflective of chronc adaptive states for 'wear & tear' of the human body
  Score: 0-5
  Higher score indicating higher allostatic load
EuroQol-5Dimension (EQ-5D) | Once - Baseline
  Investigate quality of life levels of participants
  Score: 5-likert with no problem, slight, moderate, severe and extreme in each of the dimensions plus the 0-100 VAS as a global rating of self-perceived health with higher scores indcating better health
Pittsburgh Sleep Quality Index (PSQI) | Once - Baseline
  Assess sleep quality of participants
  Score: 0-21
  Higher scores indicate worse sleep quality
Modified Baecke Physical Activity Questionnaire (MBPAQ) | Once - Baseline
  Evaluate Physical Activity levels of participants
  Score: low - moderate - high
  Higher scores indicate higher activity levels

CONTACTS AND LOCATIONS:
Overall Officials: ELENI KAPRELI, PT, PROF, Study Director — University of Thessaly

IPD SHARING:
Plan to Share IPD: Undecided